CLINICAL TRIAL: NCT04039178
Title: The Efficacy of ElectroMagnetic Field Brain Computer Interface Based Device in the Management of Acute Stroke Patients
Brief Title: Efficacy of EMF BCI Based Device on Acute Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated at the interim point due to the covid-19 pandemic, which did not allow completing full recruitment in relevant timelines
Sponsor: BrainQ Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BQ3
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Acute Stroke
Keywords: BCI; BQ; motor function; acute stroke; EMF
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blinded, sham device controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sham device appears as real device. Only randomizer which is a third party, is unblinded. First 4 patients are non randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Real BQ treatment, 40 treatments including 20 minutes of device guided functional motor tasks.
  Interventions: Device: BQ
- Control group (Sham Comparator): Sham BQ treatment, (zero intensity) 40 treatments including 20 minutes of device guided functional motor tasks.
  Interventions: Device: Sham

INTERVENTIONS:
Device: BQ — The BQ device (BrainQ Technologies Ltd., Israel), a Brain Computer Interface based stimulation device, uses machine learning tools to identify high resolution spectral patterns associated with motor functions in EEG measurements of healthy/non healthy subjects. These patterns are then translated into a tailored frequency dependent low intensity, non-invasive electro-magnetic treatment protocol.
  Other Names: Formerly VLIFE
  Arms: Treatment group
Device: Sham — Sham BQ device
  Arms: Control group

SUMMARY:
The study tests the efficacy of a non-invasive device with low intensity electromagnetic field dedicated treatment to enhance the recovery of stroke patients impaired hand motor function

DETAILED DESCRIPTION:
The study investigates the effect of BCI based stimulation device on upper limb motor function of acute stroke patients.

The BQ device (BrainQ Technologies Ltd., Israel), a Brain Computer Interface based stimulation device, uses machine learning tools to identify high resolution spectral patterns associated with motor functions in EEG measurements of healthy/non healthy subjects. These patterns are then translated into a tailored frequency dependent low intensity, non-invasive electro-magnetic treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of 1st ever ischemic stroke confirmed by imaging or 1st recurrent ischemic stroke with no previous neurological impairment in the same limb before current stroke happened
2. 72h to 15 days from stroke onset or 21 days from stroke onset in case the patient was still unstable at day 15 from stroke onset).
3. Medically stable patients
4. Age: > 18, <80 years, and independent in their daily activities before the stroke
5. Right dominant hand
6. FM >10, <45 of upper tested limb.
7. Able to sit in a chair for 70 consecutive minutes and follow three verbal instructions:

   * Bring your healthy arm to the level of your shoulder
   * Pick up this pen with your healthy hand.
   * Put your healthy hand on your waist
8. Able to understand the information provided and provide informed consent

Exclusion Criteria

1. Contraindication for performing MRI scanning
2. History of recent epileptic seizures or epilepsy and/or currently taking medication that are known to lower the seizure threshold
3. Patients with an acute problem such as active infection at the time of recruitment for research
4. Previous disease of the central nervous system
5. Damage to the joints, bones and muscles causing restriction of movement of the upper limb being tested
6. Patients known to suffer from some peripheral nerve damage of the upper limb that being tested
7. Pregnant women and women who have the ability to become pregnant unless they are on an acceptable method of contraception during the study.
8. Alcoholism or drug addiction as defined by DSM-IV within last 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment of Upper Extremity (FMA-UE) | Two months
  FMA score of upper limb, range between 0 to 66 (higher the better)

SECONDARY OUTCOMES:
ARAT | two months
  Action Research Arm test
BBT | two months
  Box and Blocks test
TMT | two months
  Trail making test
NIHSS | two months
  The national institutes of health stroke scale, a 0 to 42 scale, the higher the worse.
Promis 10 | two months
  The PROMIS Global Health short form, 10 questions questionnaire, calculated through a look up t-score table
MoCA | two months
  Montreal cognitive assessment
mRs | two months
  modified Rankin scale, a 0 to 6 scale, the higher the worse
MRI-DTI | two months
  magnetic resonance imaging, diffusion tensor imaging
brain recovery biomarkers | two months
  UCH-L1, and GFAP

CONTACTS AND LOCATIONS:
Overall Officials: Dharam P Pandey, PhD, Principal Investigator — BLK hospital , New Delhi , India
Locations (1):
- BLK super specialty hospital, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weisinger B, Pandey DP, Saver JL, Hochberg A, Bitton A, Doniger GM, Lifshitz A, Vardi O, Shohami E, Segal Y, Reznik Balter S, Djemal Kay Y, Alter A, Prasad A, Bornstein NM. Frequency-tuned electromagnetic field therapy improves post-stroke motor function: A pilot randomized controlled trial. Front Neurol. 2022 Nov 14;13:1004677. doi: 10.3389/fneur.2022.1004677. eCollection 2022. PMID 36452175